CLINICAL TRIAL: NCT01852578
Title: A Pilot Phase II Trial of Cabazitaxel in Patients With Metastatic NSCLC Progressing After Docetaxel-based Treatment
Brief Title: Cabazitaxel in Relapsed and Metastatic NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/12.02
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: NSCLC
Keywords: Metastatic NSCLC; 2nd Line; Docetaxel-based treatment; Progressed; Refractory
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel: 25 mg/m² i.v over 1 h on day 1. Cycles repeated ever 3 weeks
  Other Names: Jevtana

SUMMARY:
The investigators propose to study the single agent activity of Cabazitaxel in a Phase II trial of subjects with relapsed or refractory non-small cell lung cancer pretreated with docetaxel, given the fact of its significant activity and its acceptable toxicity profile.

DETAILED DESCRIPTION:
Non small cell lung cancer represents the second most common type of cancer in both men and women in the Western world. The availability of new active regimens in the first line setting has prompted several investigators to consider second line therapy for patients with advanced NSCLC, since a substantial percentage of patients maintain a good PS upon recurrence. On the basis of the results of phase III trials docetaxel, erlotinib, gefitinib, or pemetrexed are considered as "standard" choices for second-line therapy.

However, despite the increased availability of different drugs, NSCLC remains a devastating disease with median OS which rarely exceeds 12 months.

Preclinical data of cabazitaxel have demonstrated antitumor activity in models resistant to paclitaxel and docetaxel. In cell lines resistant to cytotoxic agents, cabazitaxel induced further tumor regression.

The recommended phase 2 doses for Cabazitaxle were 20 and 25 mg/m2. Cabazitaxel showed antitumor activity in solid tumors including docetaxel-refractory metastatic castration-resistant prostate cancer and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Cytologically or histologically documented NSCLC
* PS 0-2 (WHO scale)
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (at least one measurable lesion)
* Documented disease progression to previous treatment with docetaxel regimen in 1st or 2nd line setting assessed by Response Evaluation Criteria in Solid Tumors with at least one visceral or soft-tissue metastatic lesion.
* Brain metastases are allowed, given that are clinically stable and the patient does not present neurologic symptoms.
* Previous radiotherapy, either in the adjuvant setting or for the treatment of bone metastases, is allowed provided that the measurable lesions are outside the radiation fields. Patients who were irradiated to ≥ 40% of bone marrow are not eligible for the study.
* Patients must have a recent (within 7 days prior to treatment start) biochemical and hematogical assessment as defined by adequate bone marrow (absolute neutrophil count ≥1.5 x 109 cells/L, platelets ≥100 x 109cells/L and hemoglobin ≥9 g/dL), liver (AST & ALT ≤ 2.5x ULN, total bilirubin within normal range) and renal (serum creatinine < 1.5 x ULN). If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded) function tests
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Before patient enrollment, written informed consent must be given according to ICH/GCP and national/local regulations.

Exclusion Criteria:

* Persistence of clinically relevant treatment-related toxicities from previous chemotherapy or radiotherapy.
* Treatment with other investigational drugs or treatment in another clinical trial within the past four weeks before start of treatment or concomitantly with this trial.
* Other malignancy within the past five years other than basal cell skin cancer or carcinoma in situ of the cervix.
* Patient with reproductive potential not implementing accepted and effective method of contraception
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs or to docetaxel
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus, hypertension, heart failure ≤ NYHA II, history of myocardial infarction within the past 6 months, angina, chronic obstructive pulmonary disease (COPD), serious infections requiring systemic antibiotic therapy (e.g. antimicrobial, antifungal, antiviral)
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix A and B)
* Prior surgery, radiation, chemotherapy, within 4 weeks prior to treatment
* Active grade ≥2 peripheral neuropathy
* Active grade ≥2 stomatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Disease evaluation at Week 6

SECONDARY OUTCOMES:
Disease control rate | Disease evaluation at Week 6
  Disease control rate is defined as the proportion of patients with complete response plus partial response plus stable disease
Progression Free Survival | 1 year
Overall Survival | 1 year
Toxicity profile | Every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Athanasio Kotsakis, MD, Principal Investigator — University Hospital of Herklion
Locations (5):
- Greece (5):
  - "Ag. Georgios" General Hospital of Chania, Chania, Crete
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion, Crete
  - "IASO" General Hospital of Athens Athens, Greece, Athens
  - Air Forces Military Hospital of Athens Athens, Greece, Athens
  - "PAPAGEORGIOY" General Hospital of Thessaloniki, Thessaloniki